CLINICAL TRIAL: NCT00269893
Title: A Phase III Double-Blind, Placebo-Controlled Multicenter Study of Abciximab In Patients Undergoing High Risk Coronary Angioplasty (EPIC)
Brief Title: A Study Evaluating the Efficacy and Safety of Abciximab, an Anti-platelet Therapy, in Patients Undergoing High-risk Coronary Angioplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR006268; C0116T09 (Other: Centocor)
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Angina, Unstable; Angioplasty, Transluminal, Percutaneous Coronary
Keywords: Abciximab; Angina, unstable; Angioplasty, transluminal, Percutaneous coronary
MeSH Terms: conditions — Angina, Unstable | interventions — Abciximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive matching placebo solution bolus followed by matching placebo solution infusion up to 12 hours.
  Interventions: Drug: Placebo
- Abciximab and Placebo (Experimental): Participants will receive 0.25 milligram per kilogram (mg/kg) of body weight of abciximab (c7E3 Fab) bolus injection followed by followed by placebo solution infusion up to 12 hours.
  Interventions: Drug: Abciximab; Drug: Placebo
- Abciximab (Experimental): Participants will receive 0.25 mg/kg of body weight of abciximab bolus followed by abciximab (c7E3 Fab) infusion up to 12 hours.
  Interventions: Drug: Abciximab

INTERVENTIONS:
Drug: Abciximab — 0.25 mg/kg of body weight of abciximab either bolus or infusion.
  Other Names: c7E3 Fab
  Arms: Abciximab; Abciximab and Placebo
Drug: Placebo — Matching Placebo soulution either bolus or infusion.
  Arms: Abciximab and Placebo; Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of abciximab (an anti-platelet therapy) versus placebo in patients undergoing high risk coronary angioplasty.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter study evaluating the efficacy and safety of abciximab, an anti-platelet therapy, in patients undergoing high risk coronary angioplasty. The primary outcomes of the study include any of the following: the number of deaths from any cause, or myocardial infarctions and recurrent ischemic events requiring urgent intervention (e.g., repeat angioplasty, coronary artery bypass surgery, intracoronary stent placement, or intra-aortic balloon pump).

Patients receive an abciximab bolus, abciximab bolus plus infusion, or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for elective or urgent coronary balloon angioplasty or atherectomy with an FDA-approved device in one of the following settings: unstable angina or non-Q wave myocardial infarction, acute Q-wave myocardial infarction, or high-risk clinical/morphological characteristics

Exclusion Criteria:

* Patients with a history of hemorrhagic diathesis - Having had major surgery or clinically significant gastrointestinal or genitourinary bleeding within 6 weeks of study enrollment
* Having had a stroke within 2 years prior to enrollment or any stroke with significant residual neurological deficit
* Having occlusion of the left main coronary artery greater than 50% or a history of vasculitis
* Treated with oral anticoagulants within 7 days (unless prothrombin time is =< 1.2 times control) or intravenous dextran (before or planned for during the treatment angioplasty)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2038 (Actual)
Dates: Start 1991-11; Primary Completion 1992-11 (Actual); Study Completion 1992-11 (Actual)

PRIMARY OUTCOMES:
Any of the following within 30 days: Death from any cause; Myocardial infarction; Recurrent ischemic event requiring urgent intervention (repeat angioplasty, coronary artery bypass surgery, intracoronary stent placement, or intra-aortic balloon pump). | 30 days after angioplasty

SECONDARY OUTCOMES:
Number of participants With use of thrombolytic agent in catheterization lab | Day 1
Time spent in catheterization lab | Day 1
Number of balloon Used inflations during angioplasty | Day 1
Number of Successful Angioplasty | Day 1
Reason for Specific Mortality | Up to end of study (30 days after angioplasty)
Number of participants with late major clinical events | 30 days after angioplasty up to 6 months after angioplasty
Number of Abrupt Closure | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] EPIC Investigators. Use of a monoclonal antibody directed against the platelet glycoprotein IIb/IIIa receptor in high-risk coronary angioplasty. N Engl J Med. 1994 Apr 7;330(14):956-61. doi: 10.1056/NEJM199404073301402. PMID 8121459
- [Result] Topol EJ, Ferguson JJ, Weisman HF, Tcheng JE, Ellis SG, Kleiman NS, Ivanhoe RJ, Wang AL, Miller DP, Anderson KM, Califf RM. Long-term protection from myocardial ischemic events in a randomized trial of brief integrin beta3 blockade with percutaneous coronary intervention. EPIC Investigator Group. Evaluation of Platelet IIb/IIIa Inhibition for Prevention of Ischemic Complication. JAMA. 1997 Aug 13;278(6):479-84. doi: 10.1001/jama.278.6.479. PMID 9256222